CLINICAL TRIAL: NCT04490278
Title: COVID-19 Virtual Post Intensive Care Syndrome (CoV-PICS) Clinic: Modern, Convenient and Practical Recovery Care
Brief Title: CoV-PICS: A Virtual Post-ICU Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Chris M Palmer, Assoc Prof of Anesthesiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202007053
Record Dates: First submitted 2020-07-23; First posted 2020-07-29 (Actual); Results first posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-06

CONDITIONS: Post ICU Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with PICS (Experimental)
  Interventions: Other: Medical Record Review - Inpatient Treatment; Other: Online Questionnaires

INTERVENTIONS:
Other: Medical Record Review - Inpatient Treatment — Patient characteristics, medical history, and information regarding their inpatient treatment from the electronic medical record
Other: Online Questionnaires — Patients will complete online questionnaires related to their physical, cognitive and mental health function and inquire about current treatments. The multiprofessional CoV-PICS clinic practitioners will evaluate their responses and, combined with information obtained during their virtual visits, formulate a suggested treatment plan and needed referrals.

SUMMARY:
This is a pilot study to evaluate the feasibility of a COVID-19 virtual Post Intensive Care Syndrome (PICS) clinic (CoV-PICS). The findings from this study are the first steps in determining the feasibility and potential impact of a telehealth PICS clinic that is able to address the needs of patients with COVID-19 disease and potentially other patients that are unable to attend a brick and mortar clinic and require virtual care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* COVID-19 diagnosis with a stay in the ICU.
* A home internet connection or smartphone access, along with the ability to use them
* Missouri resident

Exclusion Criteria:

* Severe cognitive deficits or dementia prior to hospitalization
* Long-term resident of a skilled nursing facility prior to admission
* Non-English speaking (will not have an interpreter available)
* Hospice or Comfort Care at discharge
* No plans to return to some degree of independent living at the time of discharge
* Pregnant at the time of discharge
* Prisoner at the time of discharge
* Blind
* Deaf

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Palmer, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Sommer P, Lukovic E, Fagley E, Long DR, Sobol JB, Heller K, Moitra VK, Pauldine R, O'Connor MF, Shahul S, Nunnally ME, Tung A. Initial Clinical Impressions of the Critical Care of COVID-19 Patients in Seattle, New York City, and Chicago. Anesth Analg. 2020 Jul;131(1):55-60. doi: 10.1213/ANE.0000000000004830. PMID 32221172
- [Background] Rawal G, Yadav S, Kumar R. Post-intensive Care Syndrome: an Overview. J Transl Int Med. 2017 Jun 30;5(2):90-92. doi: 10.1515/jtim-2016-0016. eCollection 2017 Jun. PMID 28721340

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With PICS
Started | 20
Completed | 14
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (10.8)
No comorbidities [Count of Participants; unit: Participants] | 3
Hypertension [Count of Participants; unit: Participants] | 7
Diabetes [Count of Participants; unit: Participants] | 5
Chronic Kidney Disease [Count of Participants; unit: Participants] | 5
Asthma [Count of Participants; unit: Participants] | 2
COPD [Count of Participants; unit: Participants] | 1
Other lung disease [Count of Participants; unit: Participants] | 3
Cancer [Count of Participants; unit: Participants] | 3
Hospital length of stay (d) [Median (Inter-Quartile Range); unit: days] | 21 [8 to 26]
ICU length of stay (d) [Median (Inter-Quartile Range); unit: days] | 11 [5 to 16]
# of patients on Mechanical Ventilation (%) [Count of Participants; unit: Participants] | 7
Time on ventilator (d) [Median (Inter-Quartile Range); unit: days] | 10 [8 to 12]
# of patients on ECMO [Number; unit: # of patients on ECMO] | 0
Discharge location (%) [Count of Participants; unit: Participants]
  Home | 8
  Rehabilitation Facility | 6

OUTCOME MEASURES:

1. Primary Outcome: Acceptance With COVID-19 Virtual Post Intensive Care Syndrome (CoV-PICS) Visits - AIM
Description: Acceptability of Intervention Measure (AIM) Implementation of outcome measure. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree
Time Frame: up to 6 months after consent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 4.8 (0.31)

2. Primary Outcome: Acceptance With COVID-19 Virtual Post Intensive Care Syndrome (CoV-PICS) Visits - IAM
Description: Intervention Appropriateness Measure (IAM) Implementation of outcome measure. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree
Time Frame: up to 6 months after consent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 4.6 (0.69)

3. Primary Outcome: Acceptance With COVID-19 Virtual Post Intensive Care Syndrome (CoV-PICS) Visits - FIM
Description: Feasibility of Intervention Measure (FIM) Implementation of outcome measure. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree
Time Frame: up to 6 months after consent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 4.7 (0.55)

4. Secondary Outcome: Post Intensive Care Syndrome (PICS) Symptoms - Daily Living - Visit 1
Description: Katz Independence in Activities in Daily Living Rates daily activities by independence or dependence in completing the task (range 0-6) 0=low or patient very dependent, 6 = high or patient independent
Time Frame: Up to 6 months after consent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 5.4 (1.1)

5. Secondary Outcome: Post Intensive Care Syndrome (PICS) Symptoms - Daily Living - Visit 2
Description: as for outcome 4
Time Frame: Approximately 60 days after initial visit (scheduling dependent)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 5.8 (0.6)

6. Secondary Outcome: Post Intensive Care Syndrome (PICS) Systems - Cognitive Visit 1
Description: Montreal Cognitive Assessment (MoCA) Screening tool for mild cognitive dysfunction. Scores range from 0 to 15 with scores of 11 and above considered normal and below 11 considered cognitive impairment.
Time Frame: Up to 6 months after consent
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 11.9 (2.1)

7. Secondary Outcome: Post Intensive Care Syndrome (PICS) Systems - Cognitive Visit 2
Description: as for outcome 6
Time Frame: Approximately 60 days after initial visit (scheduling dependent)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
score on a scale | 11.1 (2.1)

8. Secondary Outcome: Post Intensive Care Syndrome (PICS) Systems - Nutrition Initial Visit
Description: Scored Patient-Generated Subjective Global Assessment (PG-SGA) The Scored PG-SGA© includes the four patient-generated historical components (Weight History, Food Intake, Symptoms and Activities and Function - also known as the PG-SGA Short Form©), the professional part, the Global Assessment, the total numerical score (0-1 No risk, 2-3 Mild risk, 4-8 Moderate risk, 9 or more High risk), and nutritional triage recommendations based on the score.
  For each component of the PG-SGA, points (0-4) are awarded depending on the impact on nutritional status. Typical scores range from 0-35 with a higher score reflecting a greater risk of malnutrition and scores ≥9 indicating a critical need for nutrition intervention and symptom management
  0-1: no intervention 2-3: patient and family education by dietician or nurse 4-8: requires intervention by dietician >9: critical need for symptom intervention
Time Frame: Up to 6 months after consent
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
Participants
  0-1 no risk | 3
  2-3 mild risk | 8
  4-8 moderate risk | 0
  9 or more severe risk | 3

9. Secondary Outcome: Post Intensive Care Syndrome (PICS) Systems - Nutrition Final Visit
Description: as for outcome 8
Time Frame: Approximately 60 days after initial visit (scheduling dependent)
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
Participants
  0-1 no risk | 3
  2-3 mild risk | 8
  4-8 moderate risk | 0
  9 or more severe risk | 3

10. Secondary Outcome: Post Intensive Care Syndrome (PICS) Symptoms - Memory
Description: ICU Memory Tool (all inclusive tool that measures multiple items as described below)
  Questionnaire of patient's memory and feelings of ICU stay. Outcomes reported as the total number of memory types per group: factual memories, memories of feelings, delusional memories, unexplained feelings of panic, intrusive memories.
Time Frame: up to 6 months after consent
Measure: Number; unit: number of memories
Arm/Group | Patients With PICS
Number analyzed (Participants) | 14
number of memories
  Number of Factual memories | 106
  Number Feelings and memories | 49
  Number of delusions | 38
  Unexplained feelings of panic | 7
  Intrusive Memories | 7

ADVERSE EVENTS:
Time Frame: 6 months after consent.
Arm/Group | Patients With PICS
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT04490278/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT04490278/ICF_001.pdf